CLINICAL TRIAL: NCT05405725
Title: A Randomized, Double-blind, Parallel-group, Active-controlled Study to Compare the Efficacy, Safety, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of Enzene Denosumab (ENZ215) and Prolia® in Postmenopausal Women With Osteoporosis
Brief Title: A Phase 3 Study to Compare Biosimilar Denosumab With Prolia®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Enzene Biosciences Ltd. (Industry)
Collaborators: Alkem Laboratories Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALK22/ENZ215-DEN2; 2021-004811-26 (EudraCT Number)
Record Dates: First submitted 2022-05-12; First posted 2022-06-06 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: The study is having two periods, in first period its parallel assignment, second period is switch over design.
Who Masked: Participant, Investigator
Masking Description: The study is having two periods, in first period its double-blind treatment period for 12 months, second period is open label switchover period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ENZ215 (Experimental): ENZ215 Injection: - 60 mg denosumab administered as a single subcutaneous injection at day 1 and at month 6
  Interventions: Biological: ENZ215
- Prolia (Active Comparator): Prolia Injection: - 60 mg denosumab administered as a single subcutaneous injection at day 1 and at month 6
  Interventions: Biological: Prolia

INTERVENTIONS:
Biological: ENZ215 — Enrolled women with postmenopausal osteoporosis receive ENZ215 (60mg)
  Arms: ENZ215
Biological: Prolia — Enrolled women with postmenopausal osteoporosis receive Prolia
  Arms: Prolia

SUMMARY:
The Study will be conducted to Compare the Efficacy, Safety, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of Enzene Denosumab (ENZ215) and Prolia® in Postmenopausal Women with Osteoporosis.

The primary goal for the study is

1. To evaluate the efficacy of ENZ215 when compared to Prolia® in patients with postmenopausal osteoporosis, in terms of change in BMD at the lumbar spine from baseline to Month 12 and
2. To compare the AUEC of sCTX levels from baseline to Month 6

DETAILED DESCRIPTION:
The study will be divided into three periods: Screening period: up to 35 days; Double-blind treatment period of 12 months; and Open-label, switch-over period of six months.

Five hundred four (504) patients (252 patients in each treatment arm) will be enrolled in this study. All eligible patients will be randomized in the double blind treatment period in a 1:1 ratio to receive either ENZ215 or Prolia® (60 mg) subcutaneously (SC) on Day 1 and Month 6. These participants will complete study at 12 months. A PK sub-study will be conducted in a subset of 120 participants with 60 participants in each arm.

A subset of 120 participants randomised to Prolia arm and who completed 12 months of the double-blind treatment period without any significant safety concerns per the Investigator's discretion will be offered to enroll in the open-label, switch-over extension period. After re-consenting for the open-label, switch-over study, the participants will be re-randomised in a 1:1 ratio to receive either ENZ215 or Prolia® (60 mg) SC at Month 12. These participants will complete the study at Month 18.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide voluntary written informed consent and able to comply with the protocol requirements
2. Postmenopausal women aged ≥ 55 and ≤ 85 years globally, except for Spain. In Spain specifically refer to the below criteria:

   1. Postmenopausal women aged ≥ 75 and ≤ 85 years with LS T-score ≤ -2.5 or
   2. Postmenopausal women aged ≥ 65 and < 75 years with LS T-score is ≤ -2.5 and a prior fragility fracture (except for hip fracture), including non-exclusionary vertebral fractures
   3. In both cases (i.e. criteria a and b), it must also be that these are women who present a contraindication for the use of bisphosphonates or who do not tolerate the oral route.
3. Body weight ≥ 50 kg and ≤ 90 kg
4. Diagnosed with osteoporosis, with absolute BMD consistent with T-scores of ≤ 2.5 and ≥ - 4.0 at the lumbar spine (L1-L4 region) as measured by dual-energy X ray absorptiometry (DXA) at screening
5. At least 5 years of postmenopausal status confirmed by follicle-stimulating hormone (FSH) levels at screening
6. At least one hip joint and two vertebrae in L1-L4 region evaluable by DXA
7. No other clinically significant medical history, vital signs, physical examination, laboratory profiles as deemed by the Investigator or designee that would pose a risk to participant safety or interfere with the study evaluation, procedures or completion

Exclusion Criteria:

1. Known hypersensitivity to denosumab or any of the excipients of the study drug
2. Known intolerance to, or malabsorption of calcium or vitamin D supplements
3. Previous exposure to Prolia® or any other denosumab biosimilar
4. Previous use of oral bisphosphonates:

   1. Used for 3 or more years cumulatively
   2. If used for < 3 years, use within the past 12 months prior to screening
5. Use of intravenous bisphosphonates within the past 5 years prior to screening. If used more than 5 years prior, patients will be excluded if cumulative use was > 3 years.
6. Use of parathyroid hormone or its derivatives, hormone replacement therapy, romosozumab, selective estrogen-receptor modulators, or tibolone or calcitonin within 12 months prior to enrollment Note: occasional use of intravaginal estrogen treatment is not exclusionary
7. Any prior use of fluoride or strontium
8. Systemic glucocorticoids (≥ 5 mg prednisone equivalent per day or cumulative dose ≥ 50 mg) for more than 10 days within 3 months prior to enrollment (topical and inhaled corticosteroids are allowed)
9. Other bone active drugs (i.e. drugs affecting bone metabolism) including heparin, anti epileptics (except for benzodiazepines and pregabalin), antidepressants such as SSRIs, SNRIs, antipsychotics, systemic ketoconazole, adrenocorticotrophic hormone (ACTH), lithium, protease inhibitors, gonadotropin releasing hormone (GnRH) agonists, or anabolic steroids within the past 3 months prior to screening or requiring treatment with these agents during the study.

   Note: Please refer to Section 6.11 for a comprehensive list of prohibited medications
10. Known sensitivity to drug products derived from mammalian cell lines such as hormones, enzymes, cytokines, bone morphogenic proteins, clotting factors, antibodies, and fusion protein therapeutics. Patients with any known hypersensitivity to complex proteins such as monoclonal antibodies will be excluded.
11. History of one severe or more than two moderate vertebral fractures per Genant classification as determined by the central reading center
12. History of hip fracture or bilateral hip replacement
13. Total hip or femoral neck T-score <-4.0
14. History and/or presence of atypical femoral fracture
15. Presence of any active healing fracture according to the Investigator's assessment
16. History of any transplant or chronic immunosuppression (including patients on immunosuppressive therapy)
17. Severe liver dysfunction (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 3 times upper limit of normal)
18. Positive testing for hepatitis B (hepatitis B virus surface antigen [HbsAg]) or hepatitis C (hepatitis C virus antibody [HCV Ab]) virology
19. Known history of human immunodeficiency virus (HIV) infection or positive serology for HIV at screening
20. Significantly impaired renal function (determined by glomerular filtration rate of < 45 mL/min/1.73 m2 by the Modification of Diet in Renal Disease (MDRD) formula, as calculated by the central laboratory) or receiving dialysis
21. Oral or dental conditions:

    1. Osteomyelitis or history and/or presence of osteonecrosis of the jaw (ONJ)
    2. Presence of risk factors for ONJ (e.g., periodontal disease, poorly fitting dentures, poor oral hygiene, invasive dental procedures such as tooth extractions within 6 months prior to screening)
    3. Active dental or jaw condition which requires oral surgery
    4. Planned invasive dental procedure
22. Major surgery within 8 weeks prior to screening or anticipated major surgery during the study
23. Clinically significant leukopenia, neutropenia, or anemia as determined by the Investigator or any other clinically significant medical condition or laboratory abnormality that, in the opinion of the Investigator, would pose a risk to patient safety or interfere with adherence to study procedures, study completion, or the interpretation of study results Note: In case of an abnormal laboratory result which in the opinion of the investigator may be an error, is borderline, or indeterminate for inclusion in the study, the investigator may consider repeating the test once in order to rule out laboratory error.
24. Patient with an active infection or history of infection as follows:

    1. Any active infection for which systemic anti-infectives were used within 4 weeks prior to randomization
    2. A serious infection defined as requiring hospitalization or intravenous anti infectives within 8 weeks prior to randomization
    3. Recurrent or chronic infections or other active infection that, in the opinion of the Investigator, might compromise the safety of the patient
25. Evidence of any of the following conditions per laboratory test results, medical history, electrocardiogram (ECG), DXA, or X-ray review:

    1. Uncontrolled hyperthyroidism or hypothyroidism Note: Clinical significance of abnormal TSH values in patients on stable replacement therapy due to hypothyroidism or on anti-thyroid medication should be assessed and discussed with the Medical Monitor.
    2. History or current hyperparathyroidism or hypoparathyroidism (intact parathyroid hormone levels not within normal range) Note: Mild secondary hyperparathyroidism in the context of vitamin D deficiency may be acceptable upon discussion with the Medical Monitor.
    3. Vitamin D deficiency defined as 25 (OH) vitamin D level < 20 ng/mL (< 50 nmol/L) Note: Patients can be enrolled if a repeat test (post supplementation) prior to enrollment shows corrected 25 (OH) vitamin D level ≥ 20 ng/mL (≥ 50 nmol/L).
    4. Current hypocalcemia (albumin-adjusted serum calcium < 8.0 mg/dL [< 2.0 mmol/L]) or hypercalcemia (albumin-adjusted serum calcium > 10.6 mg/dL [> 2.62 mmol/L])
    5. History of parathyroid surgery
    6. Any bone or metabolic disease which may affect BMD or interfere with the interpretation of the findings, e.g., osteomalacia, osteogenesis imperfecta, osteopetrosis, achondroplasia, Paget's disease, rheumatoid arthritis, ankylosing spondylitis, Cushing's disease, hyperprolactinemia, or malabsorption syndrome
    7. Any malignancy, including solid tumors, and hematologic malignancies (except basal cell carcinoma and squamous cell carcinomas of the skin, cervical, or breast ductal carcinoma in situ, that have been completely excised and are considered cured) within the last 5 years
    8. Known or suspected history of alcoholism (including heavy drinking defined as consuming more than 3 drinks on one day or more than 7 drinks per week) or substance abuse within the past 12 months prior to the first dosing that the Investigator believes would interfere with understanding or completing the study
    9. Current heavy smoking, defined as smoking 20 or more cigarettes per day.
    10. Participated in any other clinical study in last 30 days prior to screening
    11. History and/or presence of significant cardiac disease as per Investigator's discretion, including but not restricted to:

    i. History of cardiac arrhythmia or long QT syndrome or ECG abnormalities at screening indicating significant risk for safety (e.g., that required hospitalization, emergency cardioversion, or defibrillation) ii. History and/or presence of myocardial infarction within 6 months before screening iii. History and/or presence of New York Heart Association (NYHA) class III or IV heart failure
26. Suspected signs and symptoms of COVID-19/confirmed COVID-19 or with recent history of travel/contact (less than 2 weeks from screening) with any COVID-19 positive patient/isolation/quarantine

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Patients with postmenopausal osteoporosis
Enrollment: 504 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- Bulgaria (4):
  - University Hospital, Plovdiv
  - Medical Center Teodora,, Rousse
  - DCC XVII-Sofia EOOD, Sofia
  - Research Center(Medical Center Synexus Sofia EOOD), Sofia
- Czechia (8):
  - Research Center, Brno
  - G-CENTRUM Olomouc, Horní Město
  - Research Center, Pardubice
  - University Hospital., Pilsen
  - Synexus Czech, Prague
  - Clinic, Prague
  - Fakultni nemocnice v Motole, Prague
  - MEDICAL PLUS s.r.o., Uherské Hradiště
- Sydvestjysk Sygehus Esbjerg, Esbjerg, Denmark
- Lithuania (7):
  - JSC Saules seimos medicinos ce, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Kaunas City Polyclinic, Kaunas
  - Lithuanian University of Health Sciences Hospital, Kaunas
  - Republican Siauliai Hospital, Šiauliai
  - Vilnius University Hospital Santaros Klinikos, Vilnius
  - National Osteoporosis Center, Vilnius
- Poland (23):
  - Osteo-Medic S.C. A Racewicz, Bialystok
  - Szpital Uniwersytecki, Bydgoszcz
  - Centrum Medyczne Pratia Czestochowa, Częstochowa
  - Synexus Polska, Częstochowa
  - Synexus Polska, Gdansk
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Synexus Polska, Gdynia
  - Silmedic sp. z o.o.,ul. Gen. Wladyslawa Sikorskiego, Katowice
  - Synexus Polska, Katowice
  - ETG Kielce, ul. Zagorska, Kielce
  - Krakowskie Centrum Medyczne, Krakow
  - ETG Lodz, ul. Pilota Stanislawa Wigury, Lodz
  - Synexus Polska, Lodz
  - ETG Lublin, ul. Kunickiego, Lublin
  - Twoja Przychodnia Nowosolskie Centrum Medyczne,, Nowa Sól
  - Prywatna Praktyka Lekarska, Poznan
  - Synexus Polska, Poznan
  - Twoja Przychodnia PCM, Poznan
  - ETG Siedlce, Siedlce
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Synexus Polska, Warsaw
  - Synexus Polska, Wroclaw
  - Centrum Medyczne Kuba- Med, Zamość
- Serbia (4):
  - Institute for Rheumatology, Belgrade
  - Zvezdara University Medical Center, Belgrade
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
  - Clinical Hospital Centre Bezanijska Kosa, Zemun
- Hospital de La Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 504 participants were randomized in the study at 44 centers across 7 countries (Bulgaria, Czech Republic, Denmark, Lithuania, Poland, Spain and Serbia) between July 2022 and January 2023.
Pre-assignment Details: The study included a Screening Period of maximum 35 days prior to first drug (ENZ215 and Prolia) administration, a double-blind Treatment Period up to Week 52, and an open label switchover treatment period for a subset of 120 participants from Prolia group, with administration of the study drug on Day 1, Week 26, and Week 52.
Groups:
- Prolia: Prolia Injection:- 60 mg denosumab administered as a single subcutaneous injection at Day 1 and at 6 months
- Prolia + ENZ215; Prolia + Prolia: A subset of 120 patients initially randomized to Prolia® arm re-randomized in a 1:1 ratio (i.e. 60 patients in each arm) in an open-label switch-over period to receive either ENZ215 or Prolia® (60 mg) SC at Month 12 in order to assess the impact on immunogenicity and safety of switching patients from Prolia® to ENZ215.
Period: Double-blind Treatment Period
Arm/Group | ENZ215 | Prolia | Prolia + ENZ215 | Prolia + Prolia
Started | 253 | 251 | 0 | 0
Completed | 233 | 236 | 0 | 0
Not Completed | 20 | 15 | 0 | 0
Period: Open-label Switchover Period
Arm/Group | ENZ215 | Prolia | Prolia + ENZ215 | Prolia + Prolia
Started | 0 | 0 | 60 | 60
Completed (A subset of 120 patients initially randomized to Prolia® arm and completed 12 months of double blind treatment period are re-randomized in a 1:1 ratio (i.e. 60 patients in each arm) in an open-label switch-over period to receive either ENZ215 or Prolia® (60 mg) SC at Month 12 in order to assess the impact on immunogenicity and safety of switching patients from Prolia® to ENZ215.) | 0 (A subset of 120 patients initially randomized to Prolia® arm and completed 12 months of double blind treatment period are re-randomized in a 1:1 ratio (i.e. 60 patients in each arm) in an open-label switch-over period to receive either ENZ215 or Prolia® (60 mg) SC at Month 12 in order to assess the impact on immunogenicity and safety of switching patients from Prolia® to ENZ215.) | 0 (A subset of 120 patients initially randomized to Prolia® arm and completed 12 months of double blind treatment period are re-randomized in a 1:1 ratio (i.e. 60 patients in each arm) in an open-label switch-over period to receive either ENZ215 or Prolia® (60 mg) SC at Month 12 in order to assess the impact on immunogenicity and safety of switching patients from Prolia® to ENZ215.) | 60 (A subset of 120 patients initially randomized to Prolia® arm and completed 12 months of double blind treatment period are re-randomized in a 1:1 ratio (i.e. 60 patients in each arm) in an open-label switch-over period to receive either ENZ215 or Prolia® (60 mg) SC at Month 12 in order to assess the impact on immunogenicity and safety of switching patients from Prolia® to ENZ215.) | 60 (A subset of 120 patients initially randomized to Prolia® arm and completed 12 months of double blind treatment period are re-randomized in a 1:1 ratio (i.e. 60 patients in each arm) in an open-label switch-over period to receive either ENZ215 or Prolia® (60 mg) SC at Month 12 in order to assess the impact on immunogenicity and safety of switching patients from Prolia® to ENZ215.)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Postmenopausal Women with Osteoporosis aged ≥ 55 and ≤ 85 years
Groups:
- ENZ215: ENZ215 Injection:- 60 mg denosumab administered as a single subcutaneous injection once every 6 months
- Prolia: Prolia Injection:- 60 mg denosumab administered as a single subcutaneous injection at Day 1 and at month 6
- Total: Total of all reporting groups
Arm/Group | ENZ215 | Prolia | Total
Number analyzed (Participants) | 253 | 251 | 504
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 171 | 171 | 342
  >=65 years | 82 | 80 | 162
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253 | 251 | 504
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 253 | 251 | 504
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Efficacy of ENZ215 When Compared to Prolia in Patients With Postmenopausal Osteoporosis, in Terms of Change in Bone Mineral Density (BMD) at Lumbar Spine.
Description: The percentage change in BMD at lumbar spine (L1-L4 region) measured by DXA from baseline to month 12 and the mean (±SD) percentage change over time is displayed for the ITT set.
  The ITT analysis set consisted of all randomised participants who received at least one dose of study intervention in the double-blind treatment period. In the ITT analysis set, treatment was assigned based on the study intervention to which participants were randomised, regardless of which treatment they actually received.
Time Frame: Month 12
Population: The ITT analysis set consisted of all randomised participants who received at least one dose of study intervention in the double-blind treatment period. In the ITT analysis set, treatment was assigned based on the study intervention to which participants were randomised, regardless of which treatment they actually received.
Measure: Least Squares Mean (Standard Error); unit: % Change from Baseline
Groups:
- ENZ215: ENZ215 Injection:- 60 mg Denosumab (ENZ215) administered subcutaneously on day 1 and Month 6
- Prolia: Prolia Injection:- 60 mg Denosumab (Prolia) administered subcutaneously on day 1 and at month 6.
Arm/Group | ENZ215 | Prolia
Number analyzed (Participants) | 231 | 235
% Change from Baseline | 5.350 (0.3152) | 5.533 (0.3108)
Statistical Analysis 1: Comparison: ENZ215 vs Prolia; Comparison between Study Treatment Groups; Test type: Other — Analysis was performed using an ANCOVA model including treatment, age strata, previous treatment with bisphosphonate and baseline BMD value as covariates; Mean Difference (Final Values) = -0.195, 95% CI 2-sided [-0.9167 to 0.5259]

2. Primary Outcome: Area Under the Effect Curve (AUEC) of % Change From Baseline (%CfB) of Serum C-telopeptide of Type-1 Collagen (sCTX) Levels
Description: The AUEC of %CfB in sCTX of ENZ215 was assessed as part of pharmacodynamics assessment to compare with Prolia® in female participants with postmenopausal osteoporosis. This outcome measure was assessed for initial 6 months
Time Frame: Month 6
Population: The analysis was performed on the PD Set. The PD Set consisted of all participants in the Safety Set whose sCTX values were available in order to calculate PD parameter AUEC values for primary analysis and had no major protocol deviations which affected sCTX measurement.
Measure: Geometric Mean (95% Confidence Interval); unit: h*%
Groups:
- ENZ215: ENZ215 Injection:- 60 mg Denosumab (ENZ215) administered subcutaneously on day 1 and at month 6
- Prolia: Prolia Injection: - 60 mg Denosumab (Prolia) administered subcutaneously on day 1 and at Month 6.
Arm/Group | ENZ215 | Prolia
Number analyzed (Participants) | 234 | 237
h*% | 347382.787 [340087.2488 to 354834.8289] | 345858.423 [338640.7259 to 352229.9557]
Statistical Analysis 1: Comparison: ENZ215 vs Prolia; Comparison between Study Treatment Groups; Test type: Other — ANCOVA is performed on log-transformed data of AUEC0-6m of sCTX with treatment group as fixed effect, and baseline sCTX value as a covariate. Equivalence is established if 90% CIs of geometric mean ratio lies between 0.8 and 1.25; Geometric mean ratio = 1.004, 90% CI 2-sided [0.9795 to 1.0299]

3. Secondary Outcome: To Compare the Immunogenicity Potential of ENZ215 and Prolia
Description: ADAs incidence such as ADA positive, ADA negative, NAB positive, NAB negative assessed at baseline and different timepoints from 1 month to 12 months and during open-label switch over period assessed. Subjects were considered as post-treatment ADA and NAb positive if they had at least one "Positive" ADA and NAb result after the first drug exposure. Post-treatment ADA and NAb status was determined regardless of the results at pre-dose.
Time Frame: From Baseline to Month 12 for Double blind treatment period and to month 18 for Open label switchover treatment period
Population: The analysis was performed on Safety set. The Safety Set included all randomised participants who received at least one dose of study intervention. In the safety set, treatment was assigned based on the actual treatment that participants received.
Measure: Count of Participants; unit: Participants
Groups:
- ENZ215: ENZ215 Injection: - 60 mg Denosumab (ENZ215) administered subcutaneously on day 1 and at month 6
- Prolia: Prolia Injection: - 60 mg Denosumab (Prolia) administered subcutaneously on day 1and at month 6
- Prolia + ENZ215: A subset of 60 participants randomised to Prolia arm in double blind treatment arm and who completed 12 months of the double-blind treatment period without any significant safety concerns per the Investigator's discretion were enrolled in the open-label, switch-over extension period and receive ENZ215 (60 mg) SC at Month 12, these participants completed the study at Month 18.
- Prolia + Prolia: A subset of 60 participants randomised to Prolia arm in double blind treatment arm and who completed 12 months of the double-blind treatment period without any significant safety concerns per the Investigator's discretion were enrolled in the open-label, switch-over extension period and receive Prolia (60 mg) SC at Month 12, these participants completed the study at Month 18.
Arm/Group | ENZ215 | Prolia | Prolia + ENZ215 | Prolia + Prolia
Number analyzed (Participants) | 253 | 251 | 60 | 60
Participants
  ADA positive subjects | 252 | 247 | 60 | 60
  nAb positive subjects: number analyzed (Participants) | 251 | 251 | 60 | 60
  nAb positive subjects | 1 | 5 | 0 | 0
  ADA Negative | 0 | 0 | 0 | 0
  Nab Negative | 251 | 242 | 60 | 60

4. Secondary Outcome: To Compare the Pharmacokinetics of ENZ215 and Prolia
Description: Comparison of PK parameters of ENZ215 and Prolia over 12 months
Time Frame: 12 months
Population: The PK Set was a subset of Safety Set with at least one evaluable PK endpoint (Cmax or AUC0-6M) and no major protocol deviations affecting the PK parameters up to Month 12. All the protocol deviations (irrespective of major / minor protocol deviations) with action for analysis that led to exclusion from PK set were considered for exclusion from PK set in the PK analysis set derivation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- ENZ215: ENZ215 Injection: - 60 mg Denosumab (ENZ215) administered subcutaneously on day 1 at month 6
Arm/Group | ENZ215 | Prolia
Number analyzed (Participants) | 57 | 59
h*ng/mL
  AUC (0-1M): number analyzed (Participants) | 56 | 57
  AUC (0-1M) | 3220000 (40.4) | 3000000 (33.1)
  AUC (0-3M): number analyzed (Participants) | 54 | 57
  AUC (0-3M) | 7260000 (45.7) | 6450000 (35.2)
  AUC (0-6M): number analyzed (Participants) | 54 | 57
  AUC (0-6M) | 8420000 (48.0) | 7460000 (36.7)
  AUC (6-12M): number analyzed (Participants) | 29 | 23
  AUC (6-12M) | 312000 (232.1) | 301000 (130.5)

5. Secondary Outcome: Serum Procollagen Type 1 N-terminal Propeptide (sP1NP) Levels
Description: Percent change from baseline in type 1 N-terminal propeptide (sP1NP) levels at 6 months
Time Frame: Month 6
Population: The analysis was performed on PD set. The PD Set consisted of all participants in the Safety Set whose sCTX/P1NP values were available in order to calculate PD parameter AUEC values for primary analysis and had no major protocol deviations which affected sCTX or sP1NP measurement.
Measure: Mean (Standard Deviation); unit: Percentage Change from baseline
Arm/Group | ENZ215 | Prolia
Number analyzed (Participants) | 234 | 237
Percentage Change from baseline
  Month 1 (Day 15): number analyzed (Participants) | 234 | 235
  Month 1 (Day 15) | 8.3369 (19.5170) | 7.5198 (17.9673)
  Month 1 (Day 30): number analyzed (Participants) | 234 | 236
  Month 1 (Day 30) | -17.7485 (17.1910) | -18.3767 (23.4844)
  Month 3 (Day 90): number analyzed (Participants) | 233 | 236
  Month 3 (Day 90) | -75.7738 (15.4099) | -74.5419 (16.6630)
  Month 6 (Day 180): number analyzed (Participants) | 233 | 234
  Month 6 (Day 180) | -69.7567 (19.4086) | -69.1690 (22.8816)

6. Secondary Outcome: To Compare the Change in BMD at the Lumbar Spine at Month 6
Description: Percentage change in BMD at lumbar spine measured by DXA from baseline at month 6
Time Frame: Baseline to Month 6
Population: Percentage change in BMD at lumbar spine (L1-L4 region) measured by DXA from baseline to Month 6 for the ENZ215 and Prolia® treatment groups was compared in ITT set. The ITT analysis set consisted of all randomised participants who received at least one dose of study intervention in the double-blind treatment period. The number of subjects with 6 months available assessments have been presented here.
Measure: Least Squares Mean (Standard Error); unit: Percentage Change
Groups:
- Prolia: Prolia Injection: - 60 mg Denosumab (Prolia) administered subcutaneously on day 1 and month 6.
Arm/Group | ENZ215 | Prolia
Number analyzed (Participants) | 240 | 246
Percentage Change | 3.615 (0.2643) | 4.004 (0.2596)

7. Secondary Outcome: To Compare the Change in BMD at Total Hip and Femoral Neck
Description: Percentage change in BMD at total hip and femoral neck measured by DXA from baseline to Month to predefined timepoint
Time Frame: Baseline to Month 6 and Month 12
Population: The analysis was performed using ITT set. The ITT analysis set consisted of all randomised participants who received at least one dose of study intervention in the double-blind treatment period. In the ITT analysis set, treatment was assigned based on the study intervention to which participants were randomised, regardless of which treatment they actually received. BMD Data excluded from analysis due to major protocol deviation for few of the patients as defined in SAP.
Measure: Least Squares Mean (Standard Error); unit: Percentage Change
Arm/Group | ENZ215 | Prolia
Number analyzed (Participants) | 240 | 245
Percentage Change
  Month 6-BMD at Total Hip: number analyzed (Participants) | 240 | 244
  Month 6-BMD at Total Hip | 2.222 (0.2042) | 2.327 (0.2005)
  Month 6-BMD at Femoral Neck | 1.700 (0.2461) | 1.688 (0.2420)
  Month 12-BMD at Total Hip: number analyzed (Participants) | 231 | 235
  Month 12-BMD at Total Hip | 2.534 (0.2044) | 2.935 (0.2012)
  Month 12-BMD at Femoral Neck: number analyzed (Participants) | 231 | 235
  Month 12-BMD at Femoral Neck | 1.826 (0.2905) | 2.589 (0.2866)

ADVERSE EVENTS:
Time Frame: From Baseline to Month 12 for participants in main study and up to 18 months for participants in Open label switch over period
Description: Any medical condition that is present at the time that the patient is screened should be considered as baseline and not reported as an AE. However, if it deteriorates at any time during the study, it should be recorded as an AE.
  Any abnormal laboratory test results or other safety assessments (e.g., ECG, radiological scans, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the Investigator.
Groups:
- ENZ215: ENZ215 Injection: - 60 mg denosumab administered as a single subcutaneous injection once every 6 months. These participants completed the study at Month 12.
- Prolia: Prolia Injection: - 60 mg denosumab administered as a single subcutaneous injection once every 6 months. These participants completed the study at Month 12.
- Prolia + Prolia: A subset of 60 participants randomised to Prolia arm in double blind treatment arm and who completed 12 months of the double-blind treatment period without any significant safety concerns per the Investigator's discretion were enrolled in the open-label, switch-over extension period and received Prolia® (60 mg) SC at Month 12, these participants completed the study at Month 18.
Arm/Group | ENZ215 | Prolia | Prolia + ENZ215 | Prolia + Prolia
All-Cause Mortality (participants affected / at risk) | 0/253 | 1/251 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 16/253 | 15/251 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 115/253 | 122/251 | 23/60 | 23/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENZ215 (N=253) | Prolia (N=251) | Prolia + ENZ215 (N=60) | Prolia + Prolia (N=60)
Radius Fracture (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Forearm Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulna Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chromophobe renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracic radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red Blood Cell urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SAPHO Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENZ215 (N=253) | Prolia (N=251) | Prolia + ENZ215 (N=60) | Prolia + Prolia (N=60)
Hypertension (Vascular disorders) | 9 (9) | 12 (14) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 6 (6) | 6 (6) | 0 (0) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (9) | 13 (16) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 6 (6) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 5 (6) | 0 (0) | 0 (0)
Chronic Gastritis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (9) | 4 (4) | 1 (1) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (4) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 9 (13) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 6 (6) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 18 (21) | 22 (24) | 5 (6) | 5 (5)
Bronchitis (Infections and infestations) | 11 (12) | 6 (6) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 5 (5) | 12 (12) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 6 (7) | 3 (3) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 11 (13) | 16 (19) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (6) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 8 (8) | 8 (9) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 5 (5) | 6 (6) | 0 (0) | 0 (0)
Urinary Tract Infection bacterial (Infections and infestations) | 3 (4) | 5 (5) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 5 (6) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Pulpitis Dental (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Bronchitis Bacterial (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (7) | 6 (6) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lyme Disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shoulder girdle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyslipidaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharochalasis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of conjunctiva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT05405725/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT05405725/SAP_001.pdf